CLINICAL TRIAL: NCT06941376
Title: Pragmatic, Open-Label, Two-Stage, Pilot Study of Effectiveness of Immunomodulatory Medications for Patients With Relapsing Polychondritis
Brief Title: An Open-Label Study of Effectiveness of Immunomodulatory Medications for Patients With Relapsing Polychondritis
Acronym: PROSECT RP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Shubhasree Banerjee, Assistant Professor of Clinical Medicine, University of Pennsylvania
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VCRC5565
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Relapsing Polychondritis
Keywords: Relapsing Polychondritis; RP; Vasculitis; Polychondritis, relapsing
MeSH Terms: conditions — Polychondritis, Relapsing; Vasculitis | interventions — Methotrexate; Azathioprine; Adalimumab; Infliximab; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Azathioprine or Methotrexate (Experimental)
  Interventions: Drug: Methotrexate (MTX); Drug: Azathioprine (AZA)
- Adalimumab, Infliximab, or Tocilizumab (Experimental)
  Interventions: Biological: Adalimumab; Biological: Infliximab; Biological: Tocilizumab

INTERVENTIONS:
Drug: Methotrexate (MTX) — Weekly methotrexate dose of 20 mg (oral or subcutaneous).
  Arms: Azathioprine or Methotrexate
Drug: Azathioprine (AZA) — Azathioprine dose will be 2-3 mg/kg body weight per day.
  Arms: Azathioprine or Methotrexate
Biological: Adalimumab — Adalimumab dose will be 40 mg subcutaneously every 1-2 weeks
  Arms: Adalimumab, Infliximab, or Tocilizumab
Biological: Infliximab — Infliximab dose will be 5mg/kg at week 0 and week 2, and then every 4-8 weeks.
  Arms: Adalimumab, Infliximab, or Tocilizumab
Biological: Tocilizumab — Tocilizumab dose will be 162 mg subcutaneous injection every week or 4-8 mg/kg every 4 weeks
  Arms: Adalimumab, Infliximab, or Tocilizumab

SUMMARY:
Open label pragmatic two-stage non-randomized trial comparing the effectiveness of five different standard of care treatment options for patients with relapsing polychondritis (RP).

DETAILED DESCRIPTION:
Twenty eligible patients with mild to moderately active RP within 60 days prior to screening will be enrolled to the study.

Subjects will be eligible to enroll into stage 1 if they are naïve to methotrexate (MTX) or azathioprine (AZA), or having active disease on MTX or AZA for 8 weeks or less. Patients naïve to MTX and AZA will be started on MTX. AZA will be started if there is a contraindication to MTX. Patients on MTX/AZA for 8 weeks or less with active disease will be continued with the respective medication.

Patients who do not meet primary effectiveness end point in Stage 1 or develop relapse of RP or intolerance to MTX/AZA will move to Stage 2.

Patients eligible to be enrolled to Stage 2 directly

1. History of intolerance or side effects to MTX or AZA with active disease
2. Currently on MTX or AZA for at least 8 weeks or has received it within the past 60 days for at least 8 weeks and still has mild/ moderate active disease

All patients in Stage 2 will be started on Tumor necrosis factor inhibitor (TNFi) or Interleukin 6 inhibitor (IL6i). The two TNFis that will be used in the trial are adalimumab or infliximab. The choice between the 2 TNFis will be based on patients' preference/ feasibility. The IL6i in the study will be tocilizumab.

All patients will receive glucocorticoids (GC) which will be tapered to 5 mg daily by week 21 according to a standardized schedule in both stages of the trial.

ELIGIBILITY:
Inclusion Criteria:

A. ≥18 years of age

B. Must fulfill McAdam's or Damiani's or Michet's Criteria Diagnostic Criteria for Relapsing Polychondritis McAdam's Criteria (1976)

≥ 3 criteria out of 6 of the following:

1. Bilateral auricular chondritis
2. Non-erosive seronegative polyarthritis
3. Nasal chondritis
4. Ocular inflammation
5. Respiratory tract chondritis
6. Cochlear and/or vestibular dysfunction

Damiani's Criteria (1979)

1. ≥3 of McAdam's Criteria as above
2. ≥1 of McAdam's Criteria with histological confirmation of chondritis
3. ≥2 of McAdam's Criteria with positive response to glucocorticoids or dapsone

Michet's Criteria (1986)

Presence of ≥2 of the following criteria:

1. Auricular chondritis
2. Nasal chondritis
3. Laryngotracheal chondritis

Or presence of ≥1 of the above criteria and ≥2 of the following criteria

1. Seronegative inflammatory arthritis
2. Ocular inflammation
3. Hearing loss
4. Vestibular dysfunction

C. Mild to moderately active disease within 60 days prior to screening where the symptoms cannot be attributed to any cause other than RP and which, in the investigator's opinion, requires addition/ increase in prednisone dose between 20-60 mg/ day.

At the time of enrollment and during the trial, the following symptoms of active disease which will be evaluated:

1. Auricular inflammation: defined as increase/ new onset pain/ swelling/redness of external ear(s), ear canal
2. Nasal inflammation: defined as increase/ new onset pain/ swelling/redness of external nose
3. Ocular inflammation: defined as new onset/ worsening unilateral/ bilateral episcleritis/scleritis/ uveitis.
4. Inflammatory arthritis: defined as new onset/ worsening morning stiffness≥30 minutes, physician diagnosed tenderness/swelling in ≥1 joint; new onset/ worsening costochondritis.
5. Mild to moderate airway inflammation: defined as new onset/ worsening mild to moderate inflammation of upper airway diagnosed by direct laryngoscopy and attributed to RP; abnormal CT airway/ bronchoscopy showing wall thickening of airway (larynx, trachea, bronchi) and absence of severe manifestations such as new onset SGS/tracheomalacia/ bronchomalacia.
6. Sinonasal disease: defined as new onset/ increase in nasal crusting, discharge bleeding
7. Constitutional symptoms: defined as new onset/ worsening fever, unintentional weight loss of ≥ 5% of body weight, night sweats Patients must have at least 1 of the first 5 criteria within the past 60 days prior to the enrollment.

D. Willing and able to comply with treatment and follow-up procedures.

E. Both men and women of childbearing potential must be willing to use an effective means of birth control while receiving treatment throughout the study. Effective contraception methods include abstinence, oral contraceptives (birth control pills), intra-uterine-device, diaphragm, approved hormone injections, condoms, or medical sterilization.

F. Willing and able to provide written informed consent.

Exclusion Criteria:

A. Severe disease manifestations within the past 28 days, including:

1. Severe airway inflammation with supplemental oxygen requirement, tracheostomy, airway stenting, ventilation. Patients with prior history of severe airway disease, who currently have damage will be eligible if they have mild- moderate active disease within the past 60 days at the time of enrollment.
2. Central nervous system (CNS) disease (meningitis, encephalitis, optic neuritis) requiring hospitalization/ treatment with intravenous methylprednisolone/ cyclophosphamide.
3. Cardiac disease (symptomatic valve dysfunction, heart failure) requiring active treatment for heart failure/ hospitalization/ consideration for surgery.
4. Severe ophthalmologic manifestations: severe scleritis, uveitis, retinal vasculitis, optic neuritis which is imminently vision threatening.
5. Any disease manifestation considered organ/ life-threatening felt to require treatment with prednisone>60 mg/ day or IV methylprednisolone or cyclophosphamide.

B. Patients with current/ prior use of methotrexate or azathioprine will be eligible for stage 1 or stage 2 of the study depending on the duration of treatment with the non- biologic DMARD treatment.

C. Patients with exposure to biologic DMARDS will be excluded.

D. Evidence of active infection.

E. Known infection with human immunodeficiency virus (HIV), hepatitis C, or a positive hepatitis B surface antigen.

F. Patients at risk for tuberculosis (TB) defined as follows:

1. Current clinical, radiographic or laboratory evidence of active TB, even if currently being treated. Chest x-rays (posterior/anterior and lateral) obtained within the 6 months prior to screening and TB testing (IFN gamma release assay or PPD) performed in the past month prior to screening will be accepted; however, a copy of the reports must be placed in the participant binder.
2. A history of active TB unless there is documentation that the patient had received prior anti-TB treatment that was appropriate in duration and type according to local health authority guidelines.
3. Patients with a positive TB screening test indicative of latent TB will not be eligible for the study unless they: i. Have no evidence of current TB based on chest x-ray performed during the screening period and by history and physical exam, and ii. They are currently being treated for latent TB or the site has documentation of successful prior treatment of latent TB. Treatment regimens should be dictated by local guidelines as long as the treatment dose and duration meet or exceed local health authority guidelines. Patients with latent TB may be eligible for the trial prior to completion of treatment as long as they have completed at least 4 weeks of treatment and they have no evidence of current TB on chest x-ray at screening.

G. Inability to comply with study guidelines.

H. Cytopenia: platelet count <80,000/mm3, absolute neutrophil count <1500/mm3, hematocrit < 20%.

I. Other uncontrolled disease (co-morbidity) that could prevent a subject from fulfilling the study requirements or that would increase the risk of study procedures.

J. Patients who have a present malignancy or previous malignancy within the last 5 years prior to screening (except documented history of cured non-metastatic squamous or basal cell skin carcinoma or cervical carcinoma in situ). Patients who had a screening procedure that is suspicious for malignancy, and in whom the possibility of malignancy cannot be reasonably excluded following additional clinical, laboratory or other diagnostic evaluations.

K. Receipt of an investigational agent or device within 30 days prior to enrollment

L. A live vaccination < 4 weeks before enrollment

M. Presence of any of the following diseases:

1. ANCA-associated vasculitis
2. Polyarteritis nodosa
3. Giant cell arteritis
4. Takayasu's arteritis
5. Cogan's syndrome
6. Sarcoidosis
7. Kawasaki disease
8. Tuberculosis or atypical mycobacterial infections
9. Deep fungal infections
10. Lymphoma, lymphomatoid granulomatosis, or other type of malignancy that mimics vasculitis
11. Cryoglobulinemic vasculitis
12. Systemic lupus erythematosus
13. Rheumatoid arthritis
14. Overlap with other autoimmune diseases
15. Diagnosis of VEXAS syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the study drugs for the treatment of relapsing polychondritis. | 26 weeks
  The proportion of subjects in remission at week 26

SECONDARY OUTCOMES:
Physician's global assessment of response | Assessed at weeks 0, 12, and 26
  Health-related quality of life as measured using physician's global assessment scale.
Response rates for each of the study drugs | Response evaluated weeks 12 and 26
  Proportion of patient with complete response and significant response to therapy at weeks 12 and 26
Patient's global assessment of response | Assessed at weeks 0, 12, and 26
  Health-related quality of life as measured using patient's global assessment scale.
Health-related quality of life | Assessed at weeks 0, 12, and 26
  Health-related quality of life as measured using SF-36
Time to disease flare | 26 weeks
  Disease flare defined as increase on a disease activity instrument by at least 1 point
Safety of study drugs in RP | 26 weeks
  Safety of study drugs in patients with RP as assessed by reported adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Shubhasree Banerjee, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No